CLINICAL TRIAL: NCT03193918
Title: Phase I/Ib Study of Crenolanib With Ramucirumab and Paclitaxel as Second Line Therapy for Advanced Esophagogastric Adenocarcinoma
Brief Title: Study of Crenolanib With Ramucirumab and Paclitaxel for Advanced Esophagogastric Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-017
Record Dates: First submitted 2017-06-14; First posted 2017-06-21 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Esophagogastric Adenocarcinoma
MeSH Terms: interventions — crenolanib; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crenolanib combined with ramucirumab/paclitaxel (Experimental)
  Interventions: Drug: Crenolanib; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Crenolanib — Crenolanib continuously on Days 1-28 at 1 of 3 BID doses - 60 mg, 80 mg or 100 mg
Drug: Ramucirumab — Ramucirumab IV 8 mg/kg on Days 1 and 15 q28 days
Drug: Paclitaxel — Paclitaxel IV 80 mg/m2 on Days 1, 8 and 15 q28 days

SUMMARY:
This is a single-arm phase I/Ib study of crenolanib combined with ramucirumab/paclitaxel as second line therapy for patients with advanced/metastatic adenocarcinoma of the esophagus, GEJ or stomach. Patients will be enrolled in two phases; dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the esophagus, GEJ or stomach.
* Stage IV disease or locally advanced/unresectable tumors
* Prior progression on only 1 line of chemotherapy in the advanced/metastatic setting containing a fluoropyrimidine and/or platinum compound
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1

Exclusion Criteria:

* Prior treatment with a taxane is not permitted in the dose-expansion phase. Patients in the dose escalation component may have received a taxane in the peri-operative setting, provided they developed disease recurrence >6 months after the completion of this therapy
* Known pre-existing liver disease (e.g. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
* Patients with any clinically apparent ascites or who have undergone a paracentesis within 7 days of enrollment
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease
* Patients with arterial thrombotic events, such as cerebrovascular accident or myocardial infarction, within 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
MTD of oral continuous dosing of crenolanib (3 different doses) plus ramucirumab/paclitaxel in patients defined as the highest dose level in which <2 of 6 patients develop a DLT. The DLT is based on the 1st cycle adverse events. | 5 weeks
  The DLT is based on the first cycle (35 days) adverse events. If at least 2 of 3 or 2 of up to 6 patients experience a DLT at the starting dose level, then the study will be paused and the starting dose will be re-assessed. The MTD is defined as the highest dose level in which <2 of 6 patients develop a DLT. This will constitute the first part of the study which will enroll a maximum of 18 patients.
Response rate (RR) of the combination in patients will be radiographically evaluated until progressive disease (PD), intolerable toxicity, withdrawal of consent, physician's decision, death or the completion of 6 cycles. adenocarcinoma patients | Bi-monthly for up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Ku, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Moy RH, Greally M, Chou JF, Li J, Desai AM, Chalasani SB, Won E, Kelsen DP, Ilson DH, Janjigian YY, Capanu M, Ku GY. Phase I/Ib study of crenolanib with ramucirumab and paclitaxel as second-line therapy for advanced esophagogastric adenocarcinoma. Cancer Chemother Pharmacol. 2022 Feb;89(2):255-265. doi: 10.1007/s00280-021-04384-1. Epub 2022 Jan 23. PMID 35066693